CLINICAL TRIAL: NCT04194294
Title: Intravenous Lidocaine Reduces Remifentanil and Propofol Requirements Without Altering the Electrical Stapedial Reflex Threshold in Pediatric Cochlear Implants
Brief Title: Role of LIDOCAINE IN Pediatric Cochlear Implant Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wahba bakhet (Other)
Collaborators: Bahteem Specialized Hospital (Other)
Responsible Party: Sponsor-Investigator, Wahba bakhet, Lectrure of anesthesia, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LIDOCAINE-CI
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liocaine (Active Comparator): Group Lid
  Interventions: Drug: Lidocaine
- Na CL 0.9% (Active Comparator): group C
  Interventions: Other: Na CL 0.9%

INTERVENTIONS:
Drug: Lidocaine — Before induction of anesthesia; children in group LID received an iv bolus dose of LIDOCAINE 1 mg/kg over 5 minutes followed by 1 mg Kg-1 h-1 ivi until the start of skin closure.
  Other Names: Xylocaine
  Arms: Liocaine
Other: Na CL 0.9% — Before induction of anesthesia; children in group C equivalent volumes of Na Cl 0.9% over the same period instead of LIDOCAINE.
  Other Names: isotonic saline solution
  Arms: Na CL 0.9%

SUMMARY:
The stapedius reflex protects the ear from the loud noise. The measurement of the intraoperative electrically evoked stapedial reflex threshold (ESRT) during pediatric cochlear implants (CIs) is used to confirm that the implant is functioning correctly and determine the maximum comfortable level . Total intravenous anesthesia (TIVA) with propofol and remifentanil is frequently used for pediatric CIs as it does not suppress the ESRT. However, high doses of remifentanil exacerbates postoperative pain and increased opioid consumption.

DETAILED DESCRIPTION:
Total intravenous anesthesia (TIVA) with propofol and remifentanil is frequently used for pediatric CIs as it does not suppress the ESRT. However, high doses of remifentanil exacerbates postoperative pain and increased opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

ASA I and II children

Exclusion Criteria:

uncontrolled hypertension, diabetes mellitus, liver disease, kidney disease, heart disease, allergy to lidocaine

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Remifentanil consumption | at the end of the surgey
  microgram per kilogram

SECONDARY OUTCOMES:
ESRT responses | After insertion of the electrode and after reversal of any residual muscle relaxant (TOF response > 0.9),
  the surgeon assessed ESRT response at the basal, middle, and apical areas of the electrode array by visual monitoring of the stapedius muscle using direct

IPD SHARING:
Plan to Share IPD: Undecided